CLINICAL TRIAL: NCT03284762
Title: Xarelto® on Prevention of Stroke and Noncentral Nervous System systeMIc Embolism in Treatment Naïve Asian Patients With Non-valvular Atrial Fibrillation
Brief Title: Xarelto on Prevention of Stroke and Noncentral Nervous System Systemic Embolism in Treatment-naïve Asian Patients With Non-valvular Atrial Fibrillation
Acronym: XaMINA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 18981
Record Dates: First submitted 2017-09-14; First posted 2017-09-15 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment-naïve NVAF patients in Korea and Taiwan: Patients will be followed according to routine medical practice and the frequency of visits and procedures will be performed under routine conditions. NVAF: Non-valvular atrial fibrillation
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Rivaroxaban is a direct Factor Xa inhibitor. In this non-interventional setting, the prescription and dosing scheme is up to the treatment physician, however, the recommended dosing scheme is 20mg/day (once daily) or 15 mg/day (once daily) in patients with reduced renal function

SUMMARY:
The purpose of the study is to collect additional information of Xarelto treatment in routine clinical practice. Patients affected by atrial fibrillation and who will get Xarelto as a prophylactic treatment against stroke and systemic embolism (Stroke Prevention in Atrial Fibrillation) will be observed.

DETAILED DESCRIPTION:
The study takes place in Korea and Taiwan. Approximately a total of 1200 patients will be included in the study within 12 months. The observation period for each patient is 1 year from enrollment into the study, or until withdrawal of consent or lost to follow-up. Patients will be followed according to routine medical practice and the frequency of visits and procedures will be performed under routine conditions.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients aged 19 years or older (Korea) and aged 20 years or older (Taiwan)
* Diagnosis of NVAF
* Patients for whom the decision to initiate treatment with rivaroxaban is made as per physician's routine treatment practice
* Treatment naïve regarding stroke prevention for atrial fibrillation
* Signed informed consent

Exclusion Criteria:

* Contraindications for rivaroxaban according to the local market authorization/summary of product characteristics (SmPC)
* Patients participating in an investigational program with interventions outside of routine clinical practice

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from Taiwan and Korea visiting doctors in hospitals or medical practices for treatment of atrial fibrillation
Sampling Method: Probability Sample
Enrollment: 1216 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Major bleeding events, collected as Serious Adverse Events (SAEs) or non-serious Adverse Events (AEs) | Up to one year
  Major bleeding events, collected as SAEs or non-serious AEs and defined as overt bleeding associated with:
  * A fall in hemoglobin of ≥2 g/dL, or
  * A transfusion of ≥2 units of packed red blood cells or whole blood, or
  * Occurrence at a critical site (intracranial, intra-spinal, intraocular, pericardial, intra articular, intra-muscular with compartment syndrome, retroperitoneal), or
  * Death.

SECONDARY OUTCOMES:
AEs | Up to one year
  All events which do not fall under characterization of major bleeding events as explained in section "primary outcome variables"
SAEs | Up to one year
  All events which do not fall under characterization of major bleeding events as explained in section "primary outcome variables"
All-cause mortality | Up to one year
  All events which do not fall under characterization of major bleeding events as explained in section "primary outcome variables"
Non-major bleeding events | Up to one year
  All events which do not fall under characterization of major bleeding events as explained in section "primary outcome variables"
Symptomatic thromboembolic events | Up to one year
  All events which do not fall under characterization of major bleeding events as explained in section "primary outcome variables"
Start of rivaroxaban therapy and, if applicable, stop of rivaroxaban therapy | Up to one year
  Start date and stop date will be collected to receive information on drug persistence

CONTACTS AND LOCATIONS:
Locations (2):
- Different facilities, Multiple Locations, South Korea
- Different facilities, Multiple Locations, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, time point and process of data access. As such, Bayer commits to sharing upon request from qualified researcher's patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Liu PY, Choi EK, Kim TS, Kuo JY, Lee JM, On YK, Park SW, Park HW, Shin DG, Wang L, Yen HW, Lee MH; XaMINA Investigators. XaMINA: A Real-World, Prospective, Observational Study of Treatment-Naive Patients Treated with Rivaroxaban for Stroke Prevention in Atrial Fibrillation in Asia. Adv Ther. 2022 Jul;39(7):3316-3333. doi: 10.1007/s12325-022-02102-8. Epub 2022 May 26. PMID 35616848
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com